CLINICAL TRIAL: NCT02772887
Title: Phase 1 Trial Citrulline and Type 2 Diabetes in Pregnancy
Brief Title: Nutraceutical Citrulline in Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to successfully recruit study participants
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Robert Powers, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRO15090627
Record Dates: First submitted 2016-02-12; First posted 2016-05-16 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes
Keywords: pregnancy; type 2 diabetes; asymmetric dimethylarginine; L-arginine; L-citrulline; placental growth factor (PlGF); blood pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citrulline (Experimental): Oral L-citrulline, 3 grams once per day for 3 weeks.
  Interventions: Dietary Supplement: L-Citrulline
- Placebo (Placebo Comparator): Placebo, 3 grams once per day for 3 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-Citrulline — amino acid supplement
  Arms: Citrulline
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if oral of L-citrulline (3 grams/day) for 3 weeks provided in mid-pregnancy to pregnant women with type 2 diabetes will increase the plasma L-arginine/ADMA ratio, lower maternal blood pressure and increase maternal levels of placental growth factor (PlGF).

DETAILED DESCRIPTION:
The pregnancy-specific syndrome preeclampsia is a leading cause of maternal and fetal morbidity and mortality. The underlying cause of preeclampsia is unknown, however several pre-existing maternal conditions are associated with an increased risk of preeclampsia including: diabetes, hypertension, renal dysfunction, obesity and history of preeclampsia. Specifically, the risk of preeclampsia is five times greater in women with diabetes.

Several lines of evidence indicate that endothelial dysfunction is a central feature of the pathophysiology of preeclampsia. Asymmetric dimethylarginine (ADMA) is a methylated metabolite of the amino acid L-arginine and an endogenous inhibitor of nitric oxide synthase (NOS). High concentrations of ADMA contribute to endothelial dysfunction and ADMA inhibits angiogenesis and arteriogenesis, activities important in pregnancy and deficient in preeclampsia. ADMA concentrations are higher early in pregnancy among women who later develop preeclampsia. This protocol describes a randomized placebo-controlled trial of L-citrulline in 40 pregnant women with type 2 diabetes from approximately sixteen to nineteen weeks gestation, to determine whether L-citrulline supplementation increases the plasma L-arginine/ADMA ratio, lowers maternal blood pressure and increases a circulating marker of placental function (placental growth factor PLGF).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Type 2 diabetes with hemoglobin A1c <8
* Gestational age at randomization between 14 and 16 weeks based on clinical information
* Maternal age between 14 and 40 years

Exclusion Criteria:

* Chronic hypertension
* Major fetal anomaly
* Fetal demise
* Planned termination of the pregnancy
* Collagen vascular disease (autoimmune disease) on medication
* Renal disease
* Epilepsy or other seizure disorder
* Active or chronic liver disease
* Heart disease, known illicit drug or alcohol abuse during current pregnancy
* Already taking L-citrulline as a supplement (1gram/day or more)

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure | approximately 20 weeks
  research measure

SECONDARY OUTCOMES:
Placental growth factor (PlGF) | approximately 20 weeks
  quantified by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No